CLINICAL TRIAL: NCT04356235
Title: Examining and Comparing Patient Satisfaction and Long-term Cosmetic Results Achieved With Implant-based Breast Reconstruction Surgery With Submuscular Silicone Implant After Skin Sparing / Areola Sparing / Nipple Sparing Mastectomy and Contralateral Symmetrization (With Mastopexy and/or Silicone Implant and/or Ultrapro Mesh) With Unilateral Simple Mastectomies and With Bilateral Skin-sparing Mastectomies and Implant-based Immediate Breast Reconstructions. Response-adaptive Prospective Randomized, Comparative Clinical Trial
Brief Title: Examining and Comparing the Temporal Changes and Results of Cosmetic, Quality of Life and Patient Satisfaction Achieved With Immediate and Delayed-immediate Implant-based Breast Reconstruction Procedures and Contralateral Symmetrization Techniques
Status: Recruiting | Type: Observational
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Zoltan Matrai, Head of Surgical Oncology Department, National Institute of Oncology, Hungary
Other Study IDs: Ageing-NIO
Record Dates: First submitted 2020-04-12; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Mastectomy; Lymphedema; Breast Cancer; Quality of Life
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- A:Exp-impl-mastopexy: expander-silicone implant exchange and contralateral symmetrization with mastopexy and if needed with volume reduction
  Interventions: Procedure: A: expander-silicone implant exchange and contralateral symmetrization with mastopexy and if needed with volume reduction
- B: exp-impl-mastopexy+mesh: expander-silicone implant exchange with contralateral symmetrization with mastopexy and Ultrapro sling
  Interventions: Procedure: B: expander-silicone implant exchange with contralateral symmetrization with mastopexy and Ultrapro sling
- C: exp-impl-mastopexy+implant: expander-silicone implant exchange and contralateral symmetrization with mastopexy and silicone implant augmentation
  Interventions: Procedure: C: expander-silicone implant exchange and contralateral symmetrization with mastopexy and silicone implant augmentation
- D: exp-impl-mastopexy+implant+mesh: expander-silicone implant exchange and contralateral symmetrization with mastopexy and Utrapro sling and silicone implant augmentation
  Interventions: Procedure: D: expander-silicone implant exchange and contralateral symmetrization with mastopexy and Utrapro sling and silicone implant augmentation
- E: simple masectomy: unilateral simple mastectomy
  Interventions: Procedure: E: unilateral simple mastectomy
- F: bilateral exp-impl: after bilateral SSM, ASM, NSM, expander-implant exchange
  Interventions: Procedure: F: after bilateral SSM, ASM, NSM, expander-implant exchange

INTERVENTIONS:
Procedure: A: expander-silicone implant exchange and contralateral symmetrization with mastopexy and if needed with volume reduction — expander-silicone implant exchange and contralateral symmetrization with mastopexy and if needed with volume reduction
  Groups: A:Exp-impl-mastopexy
Procedure: B: expander-silicone implant exchange with contralateral symmetrization with mastopexy and Ultrapro sling — expander-silicone implant exchange with contralateral symmetrization with mastopexy and Ultrapro sling
  Groups: B: exp-impl-mastopexy+mesh
Procedure: C: expander-silicone implant exchange and contralateral symmetrization with mastopexy and silicone implant augmentation — expander-silicone implant exchange and contralateral symmetrization with mastopexy and silicone implant augmentation
  Groups: C: exp-impl-mastopexy+implant
Procedure: D: expander-silicone implant exchange and contralateral symmetrization with mastopexy and Utrapro sling and silicone implant augmentation — expander-silicone implant exchange and contralateral symmetrization with mastopexy and Utrapro sling and silicone implant augmentation
  Groups: D: exp-impl-mastopexy+implant+mesh
Procedure: E: unilateral simple mastectomy — unilateral simple mastectomy
  Groups: E: simple masectomy
Procedure: F: after bilateral SSM, ASM, NSM, expander-implant exchange — after bilateral SSM, ASM, NSM, expander-implant exchange
  Groups: F: bilateral exp-impl

SUMMARY:
This is a response-adaptive (RAR) prospective randomized study with a long-term follow-up and the aim of this clinical study is to measure with qualitative and quantitative indicators the changes in cosmetic results, quality of life and patient satisfaction after breast reconstructive surgery with silicone implant (following SSM, ASM or NSM mastectomy) and symmetrization (mastopexy and/or silicone implant and/or Ultrapro mesh sling technique) over time.

According to the hypothesis of the study, the results of implant-based breast reconstruction and symmetrization following advanced postmastectomy techniques significantly decrease over time and later results limited patient satisfaction rate.

This is mainly due to the fact that over time, the natural breast differs from the reconstructed breast with silicone implant. Because of the different biological properties (gravity results ptosis on breast with mastopexy, significant volume increasement of the breast with mastopexy due to endocrine therapy, gradually progressive capsular contracture on the tumorous side, nipple flattening, nipple tattoo fading etc.) the two sides change differently resulting in significant asymmetry and consequently could lead to decreased patient satisfaction.

The high degree of asymmetry over time (which can be similar to the difference between the result of a simple mastectomy and natural breast (control group)), may indicates additional surgeries or usage of medical devices, putting a financial burden on the patient and the health system. On the other hand, the symmetry can be achieved with bilateral skin-sparing mastectomies and implant-based immediate or delayed-immediate reconstructions is clearly better and change less with time. The mastectomy of the contralateral disease-free side is considered as an unreasonable burden for moderate risk patients.

The information such as the need for multiple surgeries, change in symmetry over time etc., should be an important part of the professional decision-making mechanism and the surgeon should inform the patient during the primer surgery. Nowadays due to the lack of evidence-based knowledge, it is not part of the patient's information and surgical planning internationally. Planning breast units, attention, capacity and financial resources must also be provided to meet the long-term needs of patients who underwent postmastectomy breast reconstruction. Simple mastectomy with an external prosthesis can be an alternative for patients with intolerable degree of asymmetry or on the contrary, the results may justify the need for bilateral mastectomy and reconstruction even in the absence of high oncological risk and for purely symmetrical and cosmetic reasons.

DETAILED DESCRIPTION:
Introduction The indication of total breast removal is primarily the part of a correct oncological therapy, but secondly the removal of the full parenchyma can be prophylactic among high risk patients with positive genetic testing. Unlike in the US, in Europe it is not yet common to perform prophylactic breast surgery on the contralateral side among average risk patients with unilateral breast cancer.

In modern breast surgery, mastectomy means the removal of the entire glandular tissue. Surgery can be done in the absence of contraindication (eg, skin infiltration, mastitis carcinomatosis), by preserving the nipple-areola complex (NAC) and the skin layer above the parenchyma (nipple-sparing mastectomy, NSM) by removal of the whole or a part of the NAC (skin-sparing mastectomy, SSM) or by removal of the nipple but with the preservation of the areola (areola-sparing mastectomy, ASM).

It is important to emphasize that similarly to the classic simplex mastectomy in the cases of SSM, ASM and NSM techniques provided by an experienced and qualified breast surgeon, the complete oncological removal of the mammary gland is done.

The essence of advanced mastectomy techniques is that they ensure the combination of radical oncological resection and immediate (immediate breast reconstruction, IBR) or delayed-immediate breast reconstructive surgery (delayed immediate breast reconstruction, D-IBR) (insertion of a tissue expander during the first operation, then as a second step replace it with a silicone implant). It avoids all the burden and negative effects of distant flap surgery, like donor scars, loss of movements etc.

One or two-step post-mastectomy breast reconstructive surgeries are mainly implant-based techniques and less commonly autologous tissue techniques like distant pedicle flaps or free flaps. The tissue expander or silicone implant is placed primarily in a submuscular position but also can be inserted in a subcutaneous position in front of the large pectoral muscle.

The coverage of the lower pole or even the entire surface of the implant may be strengthened with biological (so-called acellular dermal matrix) or synthetic materials (Ultrapro mesh) to reduce the pressure load of the implant on the preserved skin, the consequent skin perforation and so the loss of the implant.

The international literature of immediate or delayed-immediate postmastectomy breast reconstructive techniques is extensive and the correlation between these procedures and the oncological treatments (such as adjuvant radiotherapy) are well known. According to the currently available evidence, reconstructive techniques do not adversely affect oncological outcome, so these breast surgical techniques are nowadays considered standard procedures in advanced breast cancer surgery.

The immediate or delayed-immediate implant-based reconstruction of the affected breast following skin-sparing mastectomy techniques requires almost in all cases symmetrization of the contralateral breast. Symmetrization surgery involves mastopexy, volume reduction or silicone implant augmentation, or furthermore skin-sparing mastectomy with an implant-based reconstruction corresponding to the tumorous side. Symmetrization can be performed in one step with the tumorous breast surgery or more often at a deferred time.

Postmastectomy breast reconstruction surgeries are well-known as an effective rehabilitation procedures, with significant psycho-oncological benefits to patients with low complication rates and high patient satisfaction. Postmastectomy breast reconstructive surgery however require more sophisticated surgical techniques, special expertise, longer surgical time and significantly higher costs than simplex mastectomies.

The cosmetic results and patient satisfaction achieved with the immediate postmastectomy reconstructive techniques with the use of symmetrisation, are widely studied, and high, mainly in the early postoperative period.

However, the long-term results of the more and more popular and widespread usage of skin-sparing mastectomies, immediate reconstructions and symmetrization surgery and the related patient satisfaction rates have so far not or only barely been in the focus of clinical trials, so the available scientific data is severely limited. The long-term disease-free survival with multidisciplinary treatments in early stage breast cancer could raise up to 85% of patients, so knowing the long-term changes of patient satisfaction, cosmetic result and symmetry of stressful and expensive immediate or delayed-immediate postmastectomy breast reconstruction surgeries is top priority.

Aim of the study

This is a response-adaptive (RAR) prospective randomized study with a long-term follow-up and the aim of this clinical study is to measure with qualitative and quantitative indicators the changes in cosmetic results, quality of life and patient satisfaction after breast reconstructive surgery with silicone implant (following SSM, ASM or NSM mastectomy) and symmetrization (mastopexy and/or silicone implant and/or Ultrapro mesh sling technique) over time.

According to the hypothesis of the study, the results of implant-based breast reconstruction and symmetrization following advanced postmastectomy techniques significantly decrease over time and later results limited patient satisfaction rate.

This is mainly due to the fact that over time, the natural breast differs from the reconstructed breast with silicone implant. Because of the different biological properties (gravity results ptosis on breast with mastopexy, significant volume increasement of the breast with mastopexy due to endocrine therapy, gradually progressive capsular contracture on the tumorous side, nipple flattening, nipple tattoo fading etc.) the two sides change differently resulting in significant asymmetry and consequently could lead to decreased patient satisfaction.

The high degree of asymmetry over time (which can be similar to the difference between the result of a simple mastectomy and natural breast (control group)), may indicates additional surgeries or usage of medical devices, putting a financial burden on the patient and the health system. On the other hand, the symmetry can be achieve with bilateral skin-sparing mastectomies and implant-based immediate or delayed-immediate reconstructions is clearly better and change less with time. The mastectomy of the contralateral disease-free side is considered as an unreasonable burden for moderate risk patients.

The information such as the need for multiple surgeries, change in symmetry over time etc., should be an important part of the professional decision-making mechanism and the surgeon should inform the patient during the primer surgery. Nowadays due to the lack of evidence-based knowledge, it is not part of the patient's information and surgical planning internationally. Planning breast units, attention, capacity and financial resources must also be provided to meet the long-term needs of patients who underwent postmastectomy breast reconstruction. Simple mastectomy with an external prosthesis can be an alternative for patients with intolerable degree of asymmetry or on the contrary, the results may justify the need for bilateral mastectomy and reconstruction even in the absence of high oncological risk and for purely symmetrical and cosmetic reasons.

Patients and method Participation in the study is voluntary. In this response-adaptive (RAR) prospective randomized study, the used standardized surgical techniques are considered to be routine procedures in the literature and iat department as well. The oncological and reconstructive surgeries do not represent new surgical procedures for patients either in their technique nor in the indication, this prospective trial guarantee quantitative and qualitative data collection only. Applied oncological therapies are unaffected by the study and still follows the decisions of the Institute's preoperative and postoperative multidisciplinary breast cancer committee. The study does not change the complex oncological treatment in any way compared to the institute's protocol.

Response-adaptive classification in this study means that the choice of the optimal surgical technique for the patient is not affected by the clinical trial. The selection of the surgical technique is based on the decision-making models that is used for a long time, and made individually for the patient's oncological disease (eg. nipple removal), breast size and degree of ptosis (NSM vs. SSM), which is the same way as patients are treated out-of-study. The principles of selecting symmetrizational techniques are presented in the introduction. In addition, reinforcement with Ultrapro mesh is used during mastopexy when the degree of the breast ptosis is at least Grade 3 or size D according to Regnault's classification or the patient has significant pseudoptosis, so the fibrous system and the skin of the breast have a very loose structure.

Therefore, in a scientific sense, this study does not involve treatments other than routine treatment protocols.

Preoperative examinations:

* Physical examination
* Triplet examination of the breast
* Chest X-ray
* Axillary ultrasound with aspiration cytology if needed
* Required additional imaging based on the oncological staging (targeted x-ray, CT, MRI, PET)
* Routine hematological and blood test analysis
* Measurements of jugulum-nipple width, nipple midline width, and nipple inframammary-fold width
* Regnault Classification of breasts' ptosis
* Photo documentation (standard 5 directions and ap with raised arms) and the application of the BCCT.core program (regarding data protection regulations)
* Filling out the BREAST-Q questionnaire

Recorded data:

Age, body mass, height, BMI, pre-/postoperative cup sizes, presence of preoperative breast assymetry and its severity (BCCT.core software data), past history, medication, smoking habits, oncological data, cTNM, pTN, pathological data, molecular genetic subtype, neoadjuvant and adjuvant therapy, type of axillary treatment, locoregional cancer recurrance, metastasis.

Age, weight, body mass, BMI, skin type typisation (normal, atypical, seborrheals, dehidrated, hyperhydrated (oedamatic)), preoperative cup size, presence of preoperative breast assymetry and its severity (BCCT.core software data), past history, medication, smoking habits, oncological data, cTNM, pTN, pathological data, molecular genetic subtype, type of mastectomy (SM, SSM,ASM, NSM), type of primary reconstruction, neoadjuvant and adjuvant therapy, type of axillary treatment, type of delayed reconstruction, type and time of symmetrisation according to primary surgery, type of the primer surgery, bra cup size after the reconstruction and symmetrisation then measuring it yearly, the size of used silicone implant(s).

Postoperative complications were classified following Clavien-Dindo Classification.

Grade I complication (light inflammations, non-surgical haematoma or suffusion, seroma formation, partial skin/NAC loss, limited fat necrosis, SSI and lymphoedema) does not require medication or surgical treatment. Grade II complication is a Grade I complication that requires medication or surgical interaction (antibiotic therapy, resuture due SSI and multiple puncture due chronic seroma). Grade III complication requires invasive surgical action (haematoma evacuation, chronic inflammation which requires reoperation, severe fat necrosis, full skin/ NAC necrosis and wound dehiscense). Grade IV complication means temporary organ failure. Grade V complication is one that leads to death.

The following data are collected in this trial: preoperative jugulum-nipple width, nipple-midline width, nipple-IMF width, vertical and horizontal width of the areola, Regnault Classification of the breast ptosis then repeating the above measurements during the follow-up (every 6 months) with parallel photo documentation, using BCCT.core program and data recording of the BREAST-Q questionnaire and 5 point Likert-scale.

Methods Enrolled patients who require unilateral SSM, ASM, NSM, or bilateral SSM, ASM, NSM with immediate- or delayed-immediate implant based reconstruction, or only unilateral SM due oncological reason, they filled out preoperative BREAST Q questionnaire and have undergone preoperative photo documentation, BCCT.core software analysis. In case of neoadjuvant therapy, the procedure is the same and the patient selection and data recording are performed preoperatively.

The patients after oncological surgery receive adjuvant therapy based on the decision of the multidisciplinary breast cancer board of the Institute. As a second step of the reconstruction the expander-implant exchange and contralateral breast's symmetrization happens at least 6 months after the adjuvant radiotherapy, and at least 3 months after the adjuvant chemotherapy. This happens at the same time in case of bilateral skin sparing mastectomies.

Data collection: measurements of the patients, the photo documentation, filling the BCCT.core software database and the postoperative quality of life BREAST Q questionnaire made postoperatively in the 4th-6th week. Nipple reconstruction performed until the postoperative 12-16th weeks in case of SSM and ASM. During the follow-up the above mentioned measurments, photo documentation and quality of life questionnaire will be checked first in the 3rd postoperative month then after every 6 months. The follow-up lasts until the end of the 5th year. During this period, correction of the breast is not allowed. The BREAST-Q questionnaire will be checked in every 6 months and the body measurements and photo documentation happens yearly in the SM group until the end of the 5th postoperative year to evaluate the contralateral breast's ptosis.

Surgical therapy The treatment of the patients examined in the study relied on the techniques of the Breast and Sarcoma Department of the National Cancer Institute including standardized SSM, ASM and NSM, and SM in the quality of life control group. (See the detailed description of these: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 8. fejezet: Tradicional breast surgery, 8.1.1. Surgical technique of simple mastectomy and classical breast-consevring surgery; 11. fejezet Postmastectomy breast reconstruction, 11.4. Immediate breast reconstruction, 11.6. Skin-sparing and areola-sparing mastectomy, 11.7. Nipple-sparing mastectomy).

According to the valid protocol of the National Cancer Institute, the surgery of the axilla can be either sentinel lymph node biopsy or axillary lymphadenectomy/ axillary block dissection, if needed with radiotherapy of the axillary and supraclavicular region depending on the regional stage of the breast cancer. (see as well in Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 8. fejezet: Tradicional breast surgery, 8.1.2. Axillary lymph nodee dissection; 9. Sentinel lymph node biopsy in breast cancer).

See the detailed standardized techniques of immediate or delayed-immediate breast reconstruction below: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 11. fejezet Postmastectomy breast reconstruction, 11.4. Immediate breast reconstruction, 11.8. Subpectoral/subserratus implant based breast reconstruction).

For the involved patients the principles of the symmetrization surgeries at Department is standardized. To achieve the best result of symmetrisation, to built a natural shape breast choosing an optimal implant size according to the footprint width, quality, quantity and the tension of the skin at the ipsilateral tumorous breast side and volume increasement with silicone implant augmentation in submuscular position and/or volume reduction and/or mastopexy at the contralateral side.

According to the institutional practice the standardized inferior pedicle Wise technique for mastopexy from an invert-T incision is chosen. If there is an expressed taint for ptosis, in the subcutaneous layer an extra Ultrapro mesh sling is used (size of 7x15 cm) to suspened the breast. (See detailed surgical technique: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. Chapter 12. Breast shape and volume symmetrisation surgeries, nipple and areola reconstruction, 12.2. The link between removal of the breast cancer and symmetrisation.) To compare the postoperative aesthetic result of SSM and ASM, the nipple reconstruction and the NAC tattooing is obligatory. The technique of the nipple reconstruction is standardized in enrolled patients. (See detailed surgical technique: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 12. fejezet Breast shape and volume symmetrisation surgeries, nipple and areola reconstruction, 12.4.3. Techniques for reconstructing the nipple.)

Using and collecting cosmetic results The following data collected in standing position marking the midline and the IMF preoperatively then at the step of delayed reconstruction and at symmetrization: jugulum-nipple width, nipple-midline width and nipple-IMF width.

The breast ptosis examination performed according to Regnault Classification at the beginning and after symmetrization.

The primary aesthetic stage will be documented with standard photo documentation using valid BCCT.core software making it measurable which allows us to compare it. the photo documentation performed the standard way in 5 position (antero-posterior (ap), 45 degree oblique and 90 degree lateral), in ap direction both ways arms up and down with strict adherence to personal privacy policies. The patients are anonymous on the pictures without their faces, and the photo documentation performed without jewelry. The mentioned software counts measurements regarding to the photo documentation and gives a 4-point rating scale (1: excellent, 2: good, 3: acceptable, 4: non-acceptable). These numerical results can be statistically analyzed.

The quality of life is measured by BREAST-Q validated questionnaire. According to this, a score is given in a 1-100 scale measuring the variables of "satisfaction with the breast", "discomfort by radiotherapy", "psychosexual wellbeing" and "physical wellbeing".Preoperatively a preoperative questionnaire and postoperatively a postoperative questionnaire is filled. Higher rates show better quality of life. The questionnaires are filled before the procedure and after the surgery in the 3rd months and every 6th months.

Likert scale is used (1. definitely not, 2: no, 3: abstain, 4: agree, 4: definitely agree) for evaluating the subjective aesthetic outcome based on the photo documentation (preoperative, 4 weeks after delayed reconstruction with symmetrization, 3rd months, every 6 months 5 years long). Based on the photo documentation three, non-involved breast surgeons make the evaluation separately without communication. The results are collected and averaged.

Follow-up The follow-up is similar to the surgical and oncological follow-up in the National Cancer Institute, so it is not a burden for the patients The primary check-up and data registration performed preoperatively, the second check-up performed 4-6th weeks after the delayed reconstruction and symmetrization then 3rd postoperative months with photo documentation, body measurements, body mass calculation and BREAST-Q questionnaire.

After this the photo documentation, body measurements, body mass calculation and BREAST-Q questionnaire examination performed every 6 months until the 5th year.

In SM group the body measurements, photo documentation made in the 3rd months and measurements of the contralateral side and the BREAST-Q questionnaire performed every 12 months.

The bioethical background of the study It is a non-interventional clinical study is conducted by the competent regional research ethics committees in accordance with the Medical law 164 / A. § (2).

This non-interventional clinical trial is performed with the permission of the Ethical Committee of the National Cancer Institute according to the 23/2002. (V.9.) Medical Regulation.

The Researchers commit themselves to protect the patient's data, photo documentation in accordance with the WHO Good Clinical Practice ( based on the Helsinki Declaration) and the applicable provisions of the General Data Protection Regulation (GDPR) regarding the international ethical and scientific quality requirements pertaining to the design, conduct, documentation and reporting principles of tests conducted on humans.

Data collection and registration It is performed with the registration sheet for computer processing and BREAST-Q questionnaire which is an internationally validated and authorized mirror translated questionnaire. Digital photo documentation (standard 5 direction with lowered arms and ap direction with raised arms) The BCCT.core made with at least 9 megapixel photo documentation, ap and lateral directions with lowered and raised arm to calculate numerically with a validated procedure the aesthetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Under the age of 65 with uni- or bilateral primary breast cancer ( clinical Stage 0-III), needing modern skin sparing mastectomy, nipple sparing mastectomy or areola sparing mastectomy independently of the axillary surgery, having immediate or delayed-immediate implant based reconstrucion on the ipsilateral side and symmetrisation on the contralateral side ( mastopexy and/or implant based reconstruction and/or breast sling with ultrapro mesh)
* Control group: patients under 65 years with unilateral simplex mastectomy without breast reconstruction

Exclusion Criteria:

* In case the patient does not volunteer for the examination or the follow-ups
* Age above 65 years or poor general health condition, where the estimated life expectancies would be less than 2 years even without the tumorous disease
* Malignant invasive tumor in the past history (except for non-melanoma skin tumors)
* Mastectomyand reconstruction performed due pregnancy associated breast cancer
* Prior breast surgery (e.g. aesthetic surgery, mastopexy) and/or radiotherapy on the breast or in the axilla
* Malignant tumor is not removed completely with pathological examination
* Severe non-surgical (e.g. radiotherapy) complication, which could influence the aesthetic and functional results
* Autoimmune diseases
* Mastitis carcinomatosa
* Lymphangitis carcinomatosa
* Open wound therapy due SSI
* Long-term steroid usage, which changed the skin's quality and structure
* Patient under foster care, or psychically non-cooperative patient
* If breast correction performed during the 5 years follow up

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The aim of the study is to evaluate the time related cosmetic results in the subgroups of implant based postmastectomy reconstruction: mastopexy, mastopexy with Ultrapro sling technique, mastopexy with silicone implant and mastopexy with silicone implant and Ultrapro sling technique. The planned subgroups contain of 80-80 cases and the control group contains also 80 cases. Planned number of the patients (calculated patients number plus 10%): 80x6=480+ 48 cases ∑528 cases should be included.
Sampling Method: Probability Sample
Enrollment: 528 (Estimated)
Dates: Start 2020-04-27 (Estimated); Primary Completion 2022-04-10 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life: BREAST-Q validated questionnaire | up to 5 years
  Correlation analysis of quality of life achieved by various surgical techniques. The quality of life is measured by BREAST-Q validated questionnaire. According to this, we give a score in a 1-100 scale measuring the variables of "psychosexual wellbeing" and "physical wellbeing". We use preoperatively a preoperative questionnaire and postoperatively a postoperative questionnaire. Higher rates show better quality of life. The questionnaires are filled before the procedure and after the surgery 4th-6th weeks then postoperatively in the 3rd months and every 6th months
Patient satisfaction: BREAST-Q validated questionnaire | up to 5 years
  Correlation analysis of patients' satisfaction achieved by various surgical techniques. The patients' satisfaction life is measured by BREAST-Q validated questionnaire. According to this, we give a score in a 1-100 scale measuring the variables of "satisfaction with the breast", "discomfort by radiotherapy" We use preoperatively a preoperative questionnaire and postoperatively a postoperative questionnaire. Higher rates show better patients' satisfaction. The questionnaires are filled before the procedure and after the surgery 4th-6th weeks then postoperatively in the 3rd months and every 6th months.

SECONDARY OUTCOMES:
Objective cosmetic results | up to 5 years
  To exclude subjectivity, the aesthetic results were classified objectively based on photo documentation using the Breast Cancer Conservative Treatment-cosmetic results (BCCT.core) software (version 20). The photo documentation performed the standard way in 5 position (antero-posterior (ap), 45 degree oblique and 90 degree lateral), in ap direction both ways arms up and down with strict adherence to personal privacy policies. BCCT.core software provides an extensive set of automated measurements using digital marks to establish a 4-point classification scale (excellent, good, fair and poor) and the overall assessment of cosmetic outcomes. Objective aesthetic results classified as fair or poor by the BCCT.core software were considered unacceptable. These numerical results can be statistically analyzed. The results are collected and averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galimberti V, Vicini E, Corso G, Morigi C, Fontana S, Sacchini V, Veronesi P. Nipple-sparing and skin-sparing mastectomy: Review of aims, oncological safety and contraindications. Breast. 2017 Aug;34 Suppl 1(Suppl 1):S82-S84. doi: 10.1016/j.breast.2017.06.034. Epub 2017 Jun 30. PMID 28673535
- [Background] Murthy V, Chamberlain RS. Defining a place for nipple sparing mastectomy in modern breast care: an evidence based review. Breast J. 2013 Nov-Dec;19(6):571-81. doi: 10.1111/j.1524-4741.2011.01220.x. Epub 2012 Jan 29. PMID 22284266
- [Background] Weber WP, Haug M, Kurzeder C, Bjelic-Radisic V, Koller R, Reitsamer R, Fitzal F, Biazus J, Brenelli F, Urban C, Paulinelli RR, Blohmer JU, Heil J, Hoffmann J, Matrai Z, Catanuto G, Galimberti V, Gentilini O, Barry M, Hadar T, Allweis TM, Olsha O, Cardoso MJ, Gouveia PF, Rubio IT, de Boniface J, Svensjo T, Bucher S, Dubsky P, Farhadi J, Fehr MK, Fulco I, Ganz-Blattler U, Gunthert A, Harder Y, Hauser N, Kappos EA, Knauer M, Landin J, Mechera R, Meani F, Montagna G, Ritter M, Saccilotto R, Schwab FD, Steffens D, Tausch C, Zeindler J, Soysal SD, Lohsiriwat V, Kovacs T, Tansley A, Wyld L, Romics L, El-Tamer M, Pusic AL, Sacchini V, Gnant M. Oncoplastic Breast Consortium consensus conference on nipple-sparing mastectomy. Breast Cancer Res Treat. 2018 Dec;172(3):523-537. doi: 10.1007/s10549-018-4937-1. Epub 2018 Sep 4. PMID 30182349
- [Background] Rowland JH, Desmond KA, Meyerowitz BE, Belin TR, Wyatt GE, Ganz PA. Role of breast reconstructive surgery in physical and emotional outcomes among breast cancer survivors. J Natl Cancer Inst. 2000 Sep 6;92(17):1422-9. doi: 10.1093/jnci/92.17.1422. PMID 10974078
- [Background] Fang SY, Shu BC, Chang YJ. The effect of breast reconstruction surgery on body image among women after mastectomy: a meta-analysis. Breast Cancer Res Treat. 2013 Jan;137(1):13-21. doi: 10.1007/s10549-012-2349-1. Epub 2012 Dec 6. PMID 23225142
- [Background] Rosenberger WF, Sverdlov O, Hu F. Adaptive randomization for clinical trials. J Biopharm Stat. 2012;22(4):719-36. doi: 10.1080/10543406.2012.676535. PMID 22651111
- [Background] Regnault P. Breast ptosis. Definition and treatment. Clin Plast Surg. 1976 Apr;3(2):193-203. PMID 1261176
- [Background] Cardoso JS, Cardoso MJ. Towards an intelligent medical system for the aesthetic evaluation of breast cancer conservative treatment. Artif Intell Med. 2007 Jun;40(2):115-26. doi: 10.1016/j.artmed.2007.02.007. Epub 2007 Apr 8. PMID 17420117
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Dikmans REG, Nene LEH, Bouman MB, de Vet HCW, Mureau MAM, Buncamper ME, Winters HAH, Ritt MJPF, Mullender MG. The Aesthetic Items Scale: A Tool for the Evaluation of Aesthetic Outcome after Breast Reconstruction. Plast Reconstr Surg Glob Open. 2017 Mar 1;5(3):e1254. doi: 10.1097/GOX.0000000000001254. eCollection 2017 Mar. PMID 28458968
- [Background] Mátrai Z, Gulyás G, Kovács T, Kásler M Principles and practice of oncoplastic breast surgery. Medicina Kiadó; 2019.
- [Background] Rizki H, Nkonde C, Ching RC, Kumiponjera D, Malata CM. Plastic surgical management of the contralateral breast in post-mastectomy breast reconstruction. Int J Surg. 2013;11(9):767-72. doi: 10.1016/j.ijsu.2013.06.844. Epub 2013 Jul 8. PMID 23845265